CLINICAL TRIAL: NCT05015673
Title: A Double-blind, Placebo-controlled, Randomized, 3-period, 3-treatment Crossover Study to Evaluate the Effect of Multiple Oral Dose Administration of SEP-363856 in Male and Female Adult Subjects With Narcolepsy-cataplexy
Brief Title: This is a Study to Determine the Effect of Multiple Doses of an Investigational Drug, Taken by Mouth, in People With Narcolepsy-cataplexy. Accepting Both Males and Females Ages of 18 Years to 55 Years. This Study Will be Conducted in the US and Will Require Approximately 13 Weeks Participation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-108
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Narcolepsy-cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: Double-blind, Placebo-controlled, Randomized, 3-period, 3-treatment Crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP-363856 25mg (Experimental): SEP-363856 25 mg given orally
  Interventions: Drug: SEP363856
- SEP-363856 50mg (Experimental): SEP-363856 50mg given orally
  Interventions: Drug: SEP363856
- Placebo (Placebo Comparator): Placebo given orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP363856
  Arms: SEP-363856 25mg; SEP-363856 50mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a study to determine the effect of multiple doses of an investigational drug, taken by mouth, in people with Narcolepsy-cataplexy.

DETAILED DESCRIPTION:
This was a multi-center, double-blind, placebo-controlled, randomized, 3-way crossover study of SEP-363856 that was conducted in adult subjects with narcolepsy-cataplexy. Two oral doses of SEP-363856 (25 and 50 mg QD for 14 days) were administered and compared with matching placebo using a 6-treatment sequence, 3-period, 3-treatment, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* To qualify for participation, subjects must meet all of the following inclusion criteria:

  1. Subject must give written informed consent and privacy authorization prior to participation in the study. Female subjects of childbearing potential and male subjects must agree to contraceptive requirements outlined in the informed consent form (ICF).
  2. Subject must be willing and able to comply with the study procedures and visit schedules and must be able to follow verbal and written instructions.
  3. Male or female subject between 18 to 55 years of age, inclusive, with narcolepsy-cataplexy (confirmation of diagnosis may occur during screening period).
  4. Subject's body mass index (BMI) must be at least 16 kg/m2 but no more than 32 kg/m2
  5. Subjects on medications for cataplexy (ie, selective serotonin reuptake inhibitors [SSRIs], serotonin and norepinephrine reuptake inhibitors [SNRIs], norepinephrine reuptake inhibitors [NRIs], tricyclic antidepressants [TCAs], or Xyrem) and/or EDS associated with narcolepsy (ie, modafinil, armodafinil, or classical stimulants such as methylphenidate and amphetamine), and/or over-the-counter (OTC) medications known to affect sleep-wake functions must washout the prohibited medications during the 2 weeks (or 5 half-lives) prior to BL-1.

     • Caffeine intake should be limited to < 300 mg (including coffee, tea, and/or other caffeine-containing beverages or foods [including, but not limited to, energy drinks, sodas, and candy]) per day for 2 weeks prior to BL-1 and throughout the study (through the EOS visit).
  6. Subject must have a negative urine drug screen (UDS) for drugs of abuse at the screening visit
  7. Male subjects with female partner(s) of childbearing potential must agree to avoid fathering a child and use acceptable methods of birth control from screening until 60 days after the last study drug administration.
  8. Female subjects must have a negative serum pregnancy test at screening.
  9. Female subjects of childbearing potential must agree to avoid pregnancy and use acceptable methods of birth control from at least 60 days prior to screening and for at least 60 days after the last study drug administration.
  10. Subject must be judged to be in a condition of general good health (defined as the absence of any clinically relevant conditions or abnormalities as determined by the Investigator), based on screening medical and psychiatric history, physical examination,neurological examination, vital signs, clinical laboratory values (hematology, chemistry, urinalysis, coagulation studies, and thyroid panel), and a 12-lead ECG.
  11. Subject must be willing to stay within the clinic for the required period.
  12. Subject must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator.
  13. Subject must agree to comply with all restrictions for the required length of time
  14. Subject must routinely spend 7 to 9 hours/night in bed and not vary bedtime by more than 2 hours in a week as determined by the sleep diary.

Exclusion Criteria:

* To qualify for study participation, subjects must not meet any of the following criteria:

  1. Subject has symptoms of any sleeping disorder other than narcolepsy-cataplexy as determined by the screening sleep history form administered by site personnel.
  2. Subject is a rotating or third-shift worker, is expected to travel (eg, transcontinental flights over 2 time zones), during the course of the study, or has a lifestyle within the prior 3 months that is disruptive to establishing a normal sleep pattern.
  3. Subject does not tolerate venipuncture or has poor venous access that would cause difficulty in collecting blood samples.
  4. Subject has participated in an investigational drug study and received investigational drug within 30 days (or longer if the elimination half-life is known to be ≥ 150 hours) prior to the screening visit, or who is currently participating in another clinical study.
  5. Subject has any clinically significant unstable acute or chronic medical condition that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:

     1. Hematologic (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urologic, cardiovascular, hepatic, neurologic, or allergic disease (except for untreated, asymptomatic, seasonal allergies at the time of dosing).
     2. History of any allergic reaction to any medication.
     3. Presence or history of a medically diagnosed, clinically significant psychiatric disorder (including mental retardation).
     4. History of cancer or significant ongoing neoplasm.
     5. Disorder or history of a condition, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection, or any surgical procedure), that may interfere with drug absorption, distribution, metabolism, excretion, or gastrointestinal motility; a clinically significant abnormality of the hepatic or renal system; or a history of malabsorption.
     6. Known or suspected substance abuse/dependence within 12 months preceding Visit 1or a positive UDS for illicit substances at screening.
     7. Known or suspected excessive alcohol consumption exceeding 14 units/week (1 unit = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor) within 6 months prior to the screening visit or a positive breath alcohol test at screening.
     8. Subject has a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study or a screening 12-lead ECG demonstrating any one of the following: heart rate > 100 beats per minute (bpm), QRS > 120 msec, QTcF > 450 msec, or PR > 220 msec.
  6. Female subject who is pregnant or lactating.
  7. Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS.
  8. Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the formulation.
  9. Subject has any clinically significant abnormal laboratory values (hematology, serum chemistry, urinalysis, coagulation studies, and thyroid panel).
  10. Subject has a history of hospitalization within 45 days prior to the screening visit.
  11. Subject has a positive test for Hepatitis B surface antigen or Hepatitis C antibody at screening.
  12. Subject has a positive test for human immunodeficiency virus (HIV-1 or HIV-2) at screening, or subject is known to have tested positive for HIV.
  13. Subject has abnormal hepatic function tests (aspartate aminotransferase [AST] > 2 x upper limit of normal [ULN], alanine aminotransferase [ALT] > 2 x ULN, bilirubin > 2 x ULN) at screening.
  14. Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to the first dose of study drug; has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.
  15. Subject consumes the equivalent of more than 10 cigarettes a day or smokes/uses nicotine-containing products from the time he/she goes to bed at night to the time he/she wakes up the next morning.
  16. Subject has a history of tobacco use associated with maintaining wakefulness or uses tobacco or nicotine-containing products (including pipe, cigar, patch, chewing tobacco, spray, inhaler, gum, or e-cigarette) to stay awake.
  17. Subject has used prescription or nonprescription drugs, vitamins, or dietary or herbal supplements including enzyme-inhibiting supplements within 30 days prior to dosing or anticipates the need for any medication during their participation in this study (exception: female subjects who are taking oral, patch, or intrauterine device [IUD] hormonal contraceptives, or progestin implant or injection). Enzyme-inducing herbal supplements (eg, Metabolife™) must be discontinued 30 days prior to the first dose of study drug. Medications for stable medical conditions that, in the opinion of the Investigator will not adversely affect a subject's participation in the study, may be allowed with prior approval of the Medical Monitor.
  18. Subject previously received study drug.
  19. Subject is a staff member or the relative of a staff member
  20. Subject is, in the opinion of the Investigator, unsuitable in any other way to participate in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total number of cataplexy attacks over the 2-week treatment period as assessed by the cataplexy diary. | Baseline and Week 2
Clinical Global Impression-Improvement (CGI-I)at the end of the 2-week treatment period to assess change in narcolepsy-cataplexy symptoms | Week 2
  The CGI-I scale is a standard 7-point scales that requires the clinician and subject, respectively, to assess how much the subject's overall narcolepsy-cataplexy symptoms improved or worsened by the end of the 2-week treatment period compared to baseline.

SECONDARY OUTCOMES:
Change from baseline in Electromyogram (EDS )at the end of the 2-week treatment period as assessed by the Mean sleep latency (mSL) from the Multiple Sleep Latency Test (MSLT). | Baseline and Week 2
Change from baseline in Excessive day time sleepiness (EDS) at the end of the 2-week treatment period as assessed by the Epworth Sleepiness Scale ( ESS). | Baseline and Week 2
  The ESS is a self-administered questionnaire that provides subjective measure of a subject's general level of daytime sleepiness. The ESS consists of 8 items, which are rated from 0 ("would never doze") to 3 ("high chance of dozing").
Change from baseline at Nights 1, 13, 30, and 47 for the following sleep architecture parameters as assessed by Nocturnal polysomnography (NPSG) | Baseline, Night 1, Night 13, Night 30, and Night 47
  * Latency to Rapid Eye Movement (REM) sleep, REM time (total minutes of REM sleep), REM percent (REM time as a percent of Total Sleep Time [TST]), and REM density (number of 3-second units per 30-second epoch with at least 1 REM).
  * Latency to persistent sleep (LPS), TST, wake after sleep onset (WASO), and number of awakenings.
  * NREM sleep stages N1, N2, and N3 time (total minutes in each stage) and percent (time in each stage as a percent of TST)
Frequency of subjects with suicidal ideation or suicidal behavior using the Columbia-Suicide Severity Rating Scale (C-SSRS) at baseline and each postbaseline visit | Week 2
  The C-SSRS is a tool designed to systematically assess and track suicidal adverse events (suicidal behavior and suicidal ideation)
Treatment-emergent adverse events, serious adverse events, concomitant medications, and change from baseline and results at each postbaseline visit in clinical evaluations | From screening to the end-of-study, an average of 90 days
  Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), concomitant medications, and change from baseline and results at each postbaseline visit in clinical evaluations (vital signs, clinical laboratory tests [hematology, serum chemistry, urinalysis, coagulation panel, and thyroid panel], and 12-lead ECGs).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - SDS Clinical Trials, Inc., Orange, California
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - Todd Swick, MD PA, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Szabo ST, Hopkins SC, Lew R, Loebel A, Roth T, Koblan KS. A multicenter, double-blind, placebo-controlled, randomized, Phase 1b crossover trial comparing two doses of ulotaront with placebo in the treatment of narcolepsy-cataplexy. Sleep Med. 2023 Jul;107:202-211. doi: 10.1016/j.sleep.2023.04.019. Epub 2023 Apr 28. PMID 37209427